CLINICAL TRIAL: NCT01054846
Title: The Impact of Helmet Use in Preschool Children From Low-income Families in Northeastern Indiana
Brief Title: Impact of Helmet Use in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parkview Hospital, Indiana (Other)
Responsible Party: Principal Investigator, Thein H Zhu, Trauma Epidemiologist, Parkview Hospital, Indiana
Organization: Parkview Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Parkview - 001
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Results first posted 2016-11-18 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Head Injuries; Facial Injuries
Keywords: Bicycle helmet
MeSH Terms: conditions — Craniocerebral Trauma; Facial Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Helmet and helmet education (Experimental): Each participant preschool child received a free bicycle Bell helmet, manufactured by Bell Sports Inc., Rantoul IL, USA. In addition, classroom bicycle helmet education was provided to all participant children and their caregivers, consisting of a video on rules of biking and the importance of proper helmet use and a classroom melon drop demonstration with and without a helmet to participants and their caregivers.
  Interventions: Other: Bicycle helmet from Bell Sports Inc.
- Helmet education (Active Comparator): Each child did not receive a bicycle Bell helmet but the child and his/her caregiver was given bicycle helmet education package as above.
  Interventions: Other: Bicycle helmet education only

INTERVENTIONS:
Other: Bicycle helmet from Bell Sports Inc. — As described under the respective arm
  Other Names: Bell bicycle helmets
  Arms: Helmet and helmet education
Other: Bicycle helmet education only — As described under the respective arm
  Other Names: Bicycle helmet education
  Arms: Helmet education

SUMMARY:
* To test the hypothesis if provision of helmet education and free helmet distribution will significantly increase helmet use in preschool children of low-income families compared to those children receiving helmet education without free helmet distribution;
* To test the hypothesis if helmet users in preschool children will significantly reduce head and facial injuries compared to those non-helmet users

DETAILED DESCRIPTION:
Current literature review shows that there were no definite prospective research studies that indicate the effectiveness of helmet promotion and wearing in injury prevention/reduction particularly to head and facial injuries among preschool children of low-income families.

The magnitude and seriousness of the injury problem in these children in the community could be high. Many injuries may occur that are not treated in emergency departments. Even the occurrence of a minor injury in the face is undesirable. These ages are learning periods to ride, are liable to fall, and are prone to injuries by using, not only, bicycles but also tricycles, scooters, roller skates/roller blades and other riding toys (vehicles).

ELIGIBILITY:
Inclusion Criteria:

* Age 3-5 year olds and their siblings, registered at the Community Action of Northeast Indiana (CANI) Head Start Program
* The child must possess a bicycle or a riding toy to ride
* The child's caregiver speaks English or Spanish

Exclusion Criteria:

* Age less than two or greater than 5-year olds
* 3-5 year old children that do not own a bicycle or a riding toy to ride
* The child's caregiver does not speak English or Spanish.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 609 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary O Aaland, MD, FACS, Study Director — Parkview Hospital Trauma Center; Thein H Zhu, MBBS, FACE, Principal Investigator — Parkview Hospital Trauma Center
Locations (1):
- Community Action of Northeast Indiana (CANI) Inc - Head Start, Fort Wayne, Indiana, United States

REFERENCES:
- [Result] Zhu TH; Aaland MO; Kerrigan C; Schiebel R; Henry H; Hollister L. Preventable head and facial injuries by providing free bicycle helmets and education to preschool children in a head start program. Health 2011 3(11):689-97
- See also: Result Publication link — http://file.scirp.org/pdf/Health20111100001_27944712.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 609 participants were enrolled in the study and 2 were later known that they did not meet study inclusion criteria.
Pre-assignment Details: Although 285 received Helmet Education only, 68 participants had prior helmet ownership and therefore were considered for further analysis.
Period: Overall Study
Arm/Group | Helmet and Helmet Education | Helmet Education
Started | 322 | 68
Completed | 246 | 51
Not Completed | 76 | 17
Not completed — Lost to Follow-up | 76 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Helmet and Helmet Education | Helmet Education | Total
Number analyzed (Participants) | 322 | 68 | 390
Age, Customized [Count of Participants; unit: Participants]
  3 years | 87 | 12 | 99
  4 years | 125 | 33 | 158
  5 years | 110 | 23 | 133
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 38 | 199
  Male | 161 | 30 | 191

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Wearing Helmet
Time Frame: Baseline (Survey 1) and 5 months (Survey 2)
Population: Analysis reflect population that owned the helmet during each survey
Measure: Number; unit: Percentage of Participants
Arm/Group | Helmet and Helmet Education | Helmet Education
Number analyzed (Participants) | 221 | 67
Percentage of Participants
  Baseline (Survey 1, n=99, 67) | 65.6 | 49.3
  5 months (Survey 2, n=221, 45) | 80.5 | 62.2
Statistical Analysis 1: Comparison: Helmet and Helmet Education; Differences between Survey 1 and Survey 2; Test type: Superiority or Other; p < 0.01, Chi-squared; z value = 2.696
Statistical Analysis 2: Comparison: Helmet Education; Difference between Survey 1 and Survey 2; Test type: Superiority or Other; p > 0.05, Chi-squared; z value = 1.351

2. Secondary Outcome: Incidence Rate of Head and Facial Injuries by Helmet Wearing Status in Helmet Owners
Description: Number of injuries by helmet wearing status as reported
Time Frame: 5 months
Population: Analysis population includes all participants that owned a helmet and available data for this assessment
Measure: Number; unit: Injuries
Arm/Group | Helmet and Helmet Education | Helmet Education
Number analyzed (Participants) | 82 | 23
Injuries
  Helmet riders (Head injuries) | 2 | 0
  Helmet riders (Face - all portions) | 12 | 3
  Helmet riders (Face - upper/mid) | 3 | 1
  Non-Helmeted riders (Head injuries) | 8 | 2
  Non-Helmeted riders (Face - all portions) | 8 | 3
  Non-Helmeted riders (Face - upper/mid) | 3 | 1

ADVERSE EVENTS:
Description: Adverse Event data was not collected per Arm; therefore a single Arm is reported.
  Other Adverse Events were monitored for the study however that detailed information is not available, because the data is no longer accessible.
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 9/607
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Study Participants (N=607)
Falls from bicycle resulting in severe injury to seek emergency care (General disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes